CLINICAL TRIAL: NCT01065597
Title: Nonconvulsive Electrotherapy: a Proof-of-concept Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Joe Smith, Director - HRPP (W. Regenold is no longer at UMD), University of Maryland, College Park
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00040324
Record Dates: First submitted 2010-02-08; First posted 2010-02-09 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2023-06-23 (Actual); Status verified 2023-05

CONDITIONS: Depressive Disorder; Bipolar Disorder; Schizoaffective Disorder
Keywords: electroconvulsive therapy; seizure; nonconvulsive; subconvulsive; major depression; bipolar disorder
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Psychotic Disorders; Seizures; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nonconvulsive electrotherapy (Experimental): Open label single arm study of nonconvulsive electrotherapy
  Interventions: Device: Nonconvulsive electrotherapy

INTERVENTIONS:
Device: Nonconvulsive electrotherapy — An electrical stimulus will be given as in electroconvulsive therapy (ECT)using bifrontal electrode placement and a Thymatron System IV device; however, the device will be set at a lower energy level that is 12.5%(1/8) of the expected energy needed to induce a seizure rather than at an energy level that is at or above the seizure threshold.
  Other Names: Thymatron System IV device made by Somatics, LLC.

SUMMARY:
This study involves pilot testing of a modified version of a proven treatment for mental illness. The treatment, electroconvulsive therapy (ECT) is used to treat more than 100,000 Americans yearly. ECT is the most effective treatment for major depression, a disorder that affects approximately 5 to 8 percent of the adult US population yearly. It is also an effective treatment for mania and mixed mood states associated with bipolar disorder and schizoaffective disorder.

The aim of ECT is to induce a seizure, which is thought to be responsible for both its therapeutic and its adverse cognitive effects. The proposed modification consists of reducing the ECT electrical stimulus dose below the amount necessary to induce seizures so that adverse cognitive effects, such as confusion and memory problems, are minimized.

The investigators intend to determine whether ECT-related cognitive impairment can be reduced without diminishing the therapeutic effect of ECT. In addition to distressing patients, ECT-related cognitive impairment has significant public health consequences. These include increased morbidity and mortality among severely ill individuals who refuse ECT due to concern over its adverse cognitive effects as well as increased falls among the elderly receiving ECT. Elderly patients are far more likely to receive ECT and are also more vulnerable to ECT-related cognitive impairment. They often require hospitalization for ECT and a longer hospital stay with greater spacing of treatments to minimize adverse cognitive effects.

The hypothesis driving this research is that electrical brain stimulation applied in the same manner as standard ECT, but at a lower dose, can have therapeutic effects and fewer adverse cognitive effects without inducing seizures. This hypothesis is based on the following: 1) the investigators clinical experience of patients who have improved with ECT despite having only one or no seizure, 2) animal studies showing that electrical brain stimulation can induce antidepressant like effects in animals without inducing seizures, 3) reports from the 1950s that "subconvulsive" and "nonconvulsive" electrotherapy was effective for some patients, and 4) the recent approval by the US Food and Drug Administration of the use of transcranial magnetic stimulation --a technique that uses a magnet to induce an electrical current in the brain without inducing seizures--for treatment of medication resistant major depression.

The primary aim of the research is to conduct a proof of concept, open trial investigating the therapeutic efficacy and safety of nonconvulsive electrotherapy (NET). The investigators plan to enroll 16 subjects, which is the minimum number of subjects needed to show that the therapeutic effect of NET is better than would be expected of placebo. If the investigators show that the therapeutic effect of NET exceeds that expected of placebo and does not induce significant cognitive impairment, then the investigators will go on to propose a blind, randomized, controlled clinical trial that more definitively tests the investigators' hypothesis. The investigators would use the information gathered from the pilot trial to estimate the number of subjects needed to definitively test the efficacy and safety of NET.

The secondary aim of the study is to find out whether NET affects blood levels of brain-derived neurotrophic factor (BDNF). BDNF is a substance that is important to the nervous system and may be related to how treatments like ECT or possibly NET improve symptoms. The investigators would draw a blood sample before and after NET treatment to assess this.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 years and older meeting structured clinical interview for the DSM IV (SCID) criteria for unipolar major depressive disorder, bipolar disorder, or schizoaffective disorder.
2. Subjects of child-bearing potential must agree to have a pregnancy test prior to enrollment and agree to use a reliable method of birth-control during the study.
3. Willingness and ability to provide informed consent as determined by satisfactorily completing the study-specific Evaluation to Sign Consent Form Test.
4. Baseline score ≥ 16 on the 21-item version of the Hamilton Depression Rating Scale (HAMD-21) for unipolar depression, the Bipolar Depression Rating Scale (BDRS) for bipolar depression, or the Young Mania rating scale (YMRS) for mania.
5. Willingness to allow the Principal Investigator to discuss study participation with treating psychiatrist
6. Taking the same regimen of psychiatric medications with no changes for at least one month prior to NET treatment and willingness to not have any medication changes during NET treatment.
7. Currently an outpatient.
8. History of or currently refusing ECT due to experience of or anticipation of adverse effects.

Exclusion Criteria:

1. Pregnancy.
2. Use of any investigational drugs within 30 days of baseline or at any time during the study.
3. Ongoing substance abuse or dependence.
4. Current suicidal ideas.
5. Presence of any condition that would contraindicate ECT or bifrontal electrode placement.
6. Medical or neurologic condition etiologically related to mood disorder.
7. History of coronary artery disease or cardiac arrhythmia.
8. History of serious, potentially life-threatening reaction to anesthesia.
9. For individuals who need to have brain imaging, presence of metal in the body that would make a head MRI unsafe.
10. For individuals who need to have brain imaging, history of claustrophobia or anxiety associated with previous MRI.
11. Allergy or adverse reaction to methohexital or succinylcholine.
12. Epilepsy or seizure disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-05; Primary Completion 2014-03 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Background] Gersner R, Toth E, Isserles M, Zangen A. Site-specific antidepressant effects of repeated subconvulsive electrical stimulation: potential role of brain-derived neurotrophic factor. Biol Psychiatry. 2010 Jan 15;67(2):125-32. doi: 10.1016/j.biopsych.2009.09.015. PMID 19880094
- [Background] BERAN M, PERKINS JC, SCOLLON RW. Psychological studies on patients undergoing nonconvulsive electric-stimulation treatment. Am J Psychiatry. 1952 Nov;109(5):367-74. doi: 10.1176/ajp.109.5.367. No abstract available. PMID 12985996
- [Derived] Regenold WT, Noorani RJ, Piez D, Patel P. Nonconvulsive Electrotherapy for Treatment Resistant Unipolar and Bipolar Major Depressive Disorder: A Proof-of-concept Trial. Brain Stimul. 2015 Sep-Oct;8(5):855-61. doi: 10.1016/j.brs.2015.06.011. Epub 2015 Jun 26. PMID 26187603

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nonconvulsive Electrotherapy
Started | 13
Completed | 12
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nonconvulsive Electrotherapy
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Score on the 17-item Hamilton Depression Rating Scale
Description: Score range is 0 to 54 points. The higher the score, the more depressed symptoms.
Time Frame: Baseline and at the end of the NET treatment course 2-4 weeks later, depending on the number of NET treatments
Population: 2 of 13 subjects had seizures during first treatment; therefore, there are no seizure-free data for them that would qualify as nonconvulsive treatment data
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nonconvulsive Electrotherapy
Number analyzed (Participants) | 11
units on a scale | -11.6 (8.2)
Statistical Analysis 1: Comparison: Nonconvulsive Electrotherapy; Test type: Superiority or Other; p = 0.001, t-test, 2 sided; This was a paired t-test

2. Secondary Outcome: Change in Score on Mini-mental State Exam
Description: Score range is 0 to 30 points. The higher the score, the better the cognition. So a higher score means less cognitive impairment.
Time Frame: Baseline and at the end of the NET treatment course 2-4 weeks later, depending on the number of NET treatments
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nonconvulsive Electrotherapy
Number analyzed (Participants) | 11
units on a scale | 0.9 (2.2)
Statistical Analysis 1: Comparison: Nonconvulsive Electrotherapy; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; This was a paired t-test

3. Secondary Outcome: Change in Score on the Autobiographical Memory Inventory Short Form (AMI-S)
Description: The Autobiographical Memory Inventory Short Form (AMI-S ) assesses effects on retrograde memory for autobiographical information including information related to a family member, recent travel, events of last New Year's eve, events of last birthday, employment information, and events of last non-psychiatric illness and its treatment. Subjects responded to specific questions regarding these topics before and after their course of NET treatment. Subjects were scored based on the percent of responses post-NET treatment that correctly matched their responses prior to NET treatment. The score range is 0 to 100%. The higher the percent, the less impaired is the autobiographical memory.
Time Frame: Baseline and at the end of the NET treatment course 2-4 weeks later, depending on the number of NET treatments
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: % correct responses
Arm/Group | Nonconvulsive Electrotherapy
Number analyzed (Participants) | 11
% correct responses | 97 (2.2)

4. Secondary Outcome: Change in Brain-derived Neurotrophic Factor (BDNF) Blood Level
Description: Change in plasma level of BDNF in pg/ml pre and post NET treatment course.
Time Frame: Baseline and at the end of the NET treatment course 2-4 weeks later, depending on the number of NET treatments
Population: 2 subjects had a seizure during the first treatment and therefore had no seizure-free (nonconvulsive) data, and 2 subjects declined blood draw
Measure: Median (Full Range); unit: pg/ml
Arm/Group | Nonconvulsive Electrotherapy
Number analyzed (Participants) | 9
pg/ml | 22 [-104 to 208]
Statistical Analysis 1: Comparison: Nonconvulsive Electrotherapy; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 4 years
Description: Subjects each participated for 2-4 weeks over the 4 year total duration of study. Participants were queried for adverse events, defined as an unwelcome change in physical or mental status that required clinical assessment, prior to and following each treatment.
Arm/Group | Nonconvulsive Electrotherapy
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 10/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nonconvulsive Electrotherapy (N=13)
Induced seizure (Nervous system disorders) | 3 — These 3 subjects had electrically induced seizure despite aim to avoid this by using a lower dose of electricity.
Headache (Nervous system disorders) | 3
Fatigue (General disorders) | 3
Jaw pain (Musculoskeletal and connective tissue disorders) | 2
Cardiac arrhythmia (Cardiac disorders) | 1
Anxiety dream (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No